CLINICAL TRIAL: NCT00616538
Title: Prospective, Randomized, Investigator-Blind, Controlled, Pilot Study Comparing Effect of Epiceram™ Device vs Standard of Care Therapy of Mid-Strength Topical Steroid (Fluticasone Propionate 0.05%) in Treatment of Atopic Dermatitis in Pediatric Subjects
Brief Title: Epiceram™ Device Versus Mid-Strength Topical Steroid (Fluticasone Propionate 0.05%) for Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ceragenix Pharmaceuticals (Industry)
Responsible Party: Sr. Vice President, Research & Development, Ceragenix Pharmaceuticals Inc.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPI 2006-002
Record Dates: First submitted 2008-02-05; First posted 2008-02-15 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-02

CONDITIONS: Atopic Dermatitis
Keywords: Atopic; Dermatitis; eczema; skin barrier; ceramide; topical; inflamation; steroid; SCORAD; glucocorticoids; EpiCeram; Cutivate; fluticasone
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cutivate(r) (Active Comparator): Topical mid-strength steroid
  Interventions: Drug: Fluticasone Propionate 0.05%
- EpiCeram(r) (Experimental): EpiCeram(r) topical barrier repair cream.
  Interventions: Device: Epiceram(r)

INTERVENTIONS:
Device: Epiceram(r) — Topical barrier repair emulsion cream
  Arms: EpiCeram(r)
Drug: Fluticasone Propionate 0.05% — Topical mid-strength steroid
  Arms: Cutivate(r)

SUMMARY:
Novel therapies for AD that avoid immunosuppression and potential carcinogensis are needed. EpiCeram™ , a topical cream, represents a novel class of therapy for skin disorders that does not contain corticosteroids or other anti-inflammatory drugs. The objective of the present study is to demonstrate the safety and efficacy of EpiCeram ™ in the treatment of moderate to severe atopic dermatitis as compared to mid-strength topical steroid cream following twice daily dosing for four weeks in pediatric patients with AD. The potential benefit to patients lies in the potential for EpiCeram ™ to provide restoration of the normal skin barrier as shown in previous studies and eliminate or reduce the requirement for supplemental topical steroid administration.

ELIGIBILITY:
Inclusion Criteria:

* Subjects willing to provide written informed consent (i.e. assent with parental/guardian consent for ages > 7 to 18 years and parental consent for ages 6 months to 7 years) to participate in the study
* Males or Females
* Age: 6 months to 18 years
* Diagnosis of Moderate to Severe Atopic Dermatitis (AD) on the basis of criteria defined by the Rajka-Langland Severity Index

Exclusion Criteria:

* Subjects with mild AD as defined by the Rajka-Laneland Severity Index.
* Subjects having greater than 20% BSA as measured by SCORAD "Extent" (A) score (total amount of body surface area requiring application of either Cutivate® or EpiCeram® exceeds 20%)
* Subjects with unstable or uncontrolled medical conditions that could require intensive treatment during the course of the study.
* Subjects who require greater than 2mg per day of inhaled or intranasal steroids.
* Subjects who are currently participating in, or have participated in another investigational drug/device trial within the past month.
* Subjects with known allergy to or hypersensitivity to EpiCeram™ or Fluticasone or Cetaphil.
* Active infection of any type at the start of the study.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 121 (Actual)
Dates: Start 2006-12; Primary Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Change in the mean Severity Scoring for Atopic Dermatitis (SCORAD) | 4 weeks

SECONDARY OUTCOMES:
Percentage of subjects reaching clear or almost clear on Investigator's Global Assessment (IGA) | 4 weeks
Change in assessments of Pruritus and sleep habits | week 4

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Sugarman, MD, Principal Investigator — University of California, San Francisco, CA; Lawrence Parrish, MD, Principal Investigator — Medical College of Thomas Jefferson University, Philadelphia, PA